CLINICAL TRIAL: NCT01223872
Title: Childhood Cancer Survivors' Knowledge of Their Diagnosis, Treatment, and Risk of Late Effects: The Impact of Care in a Specialized Survivorship Clinic
Brief Title: Childhood Cancer Survivors' Knowledge of Diagnosis,Treatment and Risk of Late Effects: Specialized Survivorship Clinic
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: VICCREACH1038
Record Dates: First submitted 2010-10-15; First posted 2010-10-19 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Childhood Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic; Ambulatory Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Routine Patient Care
  Interventions: Other: interview
- Previously-enrolled REACH Clinic Patients
  Interventions: Other: clinic visit and interview
- New REACH Clinic Patients
  Interventions: Other: interviews and clinic visit

INTERVENTIONS:
Other: interview — * Standard Interview (2-15 years from last treatment)
  * Demographic data interview (pre-initial study interview)
  Groups: Routine Patient Care
Other: clinic visit and interview — * REACH Clinic Visit(initial or regular)
  * Post-REACH Clinic Interview (3mos from initial or regular clinic visit)
  * Demographic data interview(pre-initial study interview)
  Groups: Previously-enrolled REACH Clinic Patients
Other: interviews and clinic visit — * Pre-REACH Clinic Interview(2-15 yrs from last treatment)
  * REACH Clinic Visit(initial or regular)
  * Post-REACH Clinic Interview(1mo from initial clinic visit)
  * Post-REACH Clinic Interview(3mos from initial or regular clinic visit)
  * Demographic data interview(pre-initial study interview)
  Groups: New REACH Clinic Patients

SUMMARY:
This two-part research study will compare childhood cancer survivors receiving specialized follow-up care in the REACH for Survivorship clinic to patients receiving routine follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* Treatment for primary malignancy per risk-adapted protocol
* Age ≤ 21 years at time of diagnosis
* Currently alive without evidence of disease
* Off therapy for no more than 15 years

Exclusion Criteria:

-Patients who have received a bone marrow transplant

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Fifty new cancer patients in the REACH for Survivorship clinic, fifty returning cancer patients in the REACH for Survivorship clinic, and one hundred routine care cancer patients are expected to enroll in this study.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2010-08; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Knowledge gained by attending a multispecialty Survivorship Clinic which will be measured by comparison of self report with medical record data in both cross-sectional and longitudinal approach. | 12 months
  In addition to data from patient interviews, a review of medical records will include general patient demographic data as well as data regarding cancer diagnosis, treatment and ongoing follow-up care.

SECONDARY OUTCOMES:
Characterizing how the initial consultation in a specialized clinic impacts childhood cancer survivors' knowledge of their cancer diagnosis, treatment, and risk of late effects by comparing patient's understanding among 3 sampled timepoints. | pre-clinic and a post-clinic interviews at 1 and 3 months.
An analysis of differences in relative levels of recommended screening for late effects that childhood cancer survivors have received based on the type of their long-term follow-up care comparing medical records against Survivorship Care Plan. | 12 months
  Scored responses will allow for quantitative analysis of differences within and between the cohorts of patients
A qualitative evaluation of program feedback will serve to improve the care provided in the REACH for Survivorship clinic | 12 months
  This data will be evaluated qualitatively for trends.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States